CLINICAL TRIAL: NCT04794049
Title: Oral Lactulose is Not Inferior to The Standard Bowel Preparation Regimen for Bowel Preparation Prior Colonoscopy
Brief Title: Comparison of Oral Lactulose Versus Polyethylene Glycol for Bowel Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, ZhangXiaofeng, Director of Department of Gastroenterology, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 074-1
Record Dates: First submitted 2021-01-30; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Colon Disease
Keywords: colonoscopy; bowel preparation
MeSH Terms: conditions — Colonic Diseases | interventions — Lactulose; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment cohort (Experimental): 4-6 hours before colonoscopy, patients in experiment cohort began to drink the first 150ml lactulose and half hour later, drink other 150ml lactulose dissolved in 1.5 L of water at a rate of 250ml every 15 minutes.
  Interventions: Drug: Lactulose
- Control cohort (Active Comparator): The participants in control cohort began to drink the first 2 L of PEG at 7:00-9 PM on the day before colonoscopy at a rate of 250 mL every 15 minutes. On the day of the procedure, patients took the remaining 2 L 4-6 hours before colonoscopy.
  Interventions: Drug: Polyethylene Glycol (PEG)

INTERVENTIONS:
Drug: Lactulose — In experiment cohort, patients do not use standard bowel preparation regimen, they totally drink 300ml lactulose.
  Arms: Experiment cohort
Drug: Polyethylene Glycol (PEG) — In control cohort, patients use the standard split-dose bowel preparation regimen,
  Arms: Control cohort

SUMMARY:
Adequate quality of bowel preparation(BP) is essential for colonoscopy. Several guidelines recommend that split-dose of 4L PEG should be used as a standard regime for BP. However, the high-volume PEG caused lower compliance to the regime and increased cost.

Oral lactulose is a treatment for constipation. It tastes sweet and has no obvious gastrointestinal side effects. Previous study shows 200ml lactulose oral solution plus 2L water has been proven superior BP compared to 2L PEG. However, there is a lack of research describing bowel cleansing and colonoscopy outcomes using lactulose oral solution compared with the standard split dose of 4L PEG. Here we compared the use of a lactulose oral solution (300ml+1.5 L) with a PEG formulation (2 L) for colonoscopy preparation using the following metrics: quality of cleansing, colonoscopy outcomes, patient/physician satisfaction, and patient tolerability.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 patients with intact colon and rectum

Exclusion Criteria:

* prior finding of severe colorectal stricture
* without the requirement of reaching cecum
* suspected colonic stricture or perforation
* use of prokinetic agents or purgatives within 7 days
* toxic colitis or megacolon
* pregnant women
* hemodynamically unstable
* patients who cannot give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation | 2 hours
  Boston bowel preparation score (BBPS)：cleanliness of each part of the colon: 0=unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared; 1=portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen because of staining, residual stool, and/or opaque liquid; 2=minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well; 3=entire mucosa of colon segment seen well with no residual staining, small fragments of stool, or opaque liquid.

SECONDARY OUTCOMES:
Adverse events | 2 hours
Willingness to repeat bowel preparation (BP) | 2 hours
  We will ask patients in the form of questionnaire whether they are willing to repeat the same bowel preparation method if they need colonoscopy examination again.
Adenoma detection rate | 2 hours
Insertion time | 2 hours
Withdrawal time | 2 hours
Cecal intubation rate | 2 hours

IPD SHARING:
Plan to Share IPD: Yes